CLINICAL TRIAL: NCT06428968
Title: Investigating the Central and Peripheral Insulin Resistance in Individuals With Type 2 Diabetes
Brief Title: Investigating the Insulin Resistance in Individuals With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: T2DM2024
Record Dates: First submitted 2024-05-07; First posted 2024-05-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
Keywords: Insulin resistance; Cognitive impairments
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual with type 2 diabetes (Experimental): Individual with type 2 diabetes
  Interventions: Drug: 160 units nasal insulin spray
- Healthy volunteers (Experimental)
  Interventions: Drug: 160 units nasal insulin spray

INTERVENTIONS:
Drug: 160 units nasal insulin spray — Initially, a series of MRI scans, including high-resolution T1-weighted anatomical images, diffusion tensor imaging, resting-state functional MRI, and arterial spin labeling, will be conducted. Subsequently, 160 units of nasal insulin spray will be administered, followed by a second round of MRI scans after a 30-minute interval, encompassing high-resolution T1-weighted anatomical images, resting-state functional MRI, and arterial spin labeling.

SUMMARY:
Numerous studies have provided evidence of a correlation between Type 2 Diabetes Mellitus (T2DM) and cognitive dysfunction, specifically in the realms of complex attention, information processing, and executive function. These impairments have been observed in middle-aged and elderly individuals with T2DM, with longer diabetes duration, suboptimal glycemic control, and the presence of diabetic complications being contributing factors. Recent research in young adults and adolescents diagnosed with T2DM has revealed cognitive and brain structural alterations in this growing demographic, suggesting that early disease mechanisms, rather than solely vascular and age-related neurodegeneration, contribute to pathogenesis. However, there remains uncertainty regarding the interplay between central and peripheral insulin resistance and its impact on cognitive dysfunction in individuals with T2DM. This study aims to investigate central insulin resistance in T2DM, elucidating its association with peripheral insulin resistance and the effects on cognitive impairments.

DETAILED DESCRIPTION:
Participants screened through inclusion and exclusion criteria will accept cross-sectional evaluation. The information of demographic data, medical history, previous and current medication regimen, details of complications, and family history regarding metabolic diseases will be collected. The assessments includes physical examination, anthropometry, blood test(blood routine, liver function, renal function, blood lipids, fasting blood glucose, serum insulin，thyroid function and glycosylated hemoglobin A 1c), MRI scan( High-resolution T1-weighted Anatomical Images, Diffusion Tensor Imaging, Resting-state functional MRI and Arterial Spin Labeling) and psychiatry scales(Hamilton Depression Scale, Young Mania Rating Scale and Self-reporting Inventory-90); cognitive function will be assessed by the Measurement and Treatment Research to Improve Cognition in Schizophrenia(MATRICS) Consensus Cognitive Battery; biological samples also will be collected and stored to explore related mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnostic criteria for Type 2 diabetes: typical symptoms of diabetes plus random blood glucose level of ≥11.1 mmol/l, or fasting blood glucose level of ≥7.0 mmol/l, or 2-hour post-OGTT (Oral Glucose Tolerance Test) blood glucose level of ≥11.1 mmol/l, or HbA1c level of ≥6.5%; for those without typical symptoms of diabetes, re-examination on a different day is required for confirmation.

Exclusion Criteria:

* Having history of substance dependence or abuse or whose symptoms are caused by diagnosable mental disorders;
* Having history of traumatic brain injury, seizures or other known neurological or organic diseases of the central nervous system;
* Having current suicidal or homicidal thoughts or any safety concern by research staff that cannot be manage in an inpatient setting;
* Taking drugs that could affect cognitive function.
* The routine blood tests showing significant abnormal renal, liver function or other somatic disease.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The difference of changes of brain cerebral blood flow by arterial spin labeling between type 2 diabetes and healthy volunteers. | Baseline
  Whole brain cerebral blood flow (CBF) will be recorded by arterial spin labeling (ASL). the changes in CBF (c-CBF) before and after the application of 160 units nasal insulin spray of interventional participants will be calculated. The c-CBF is an index of central insulin response.
The difference of the level of insulin signaling in Extracellular Vesicles of neuronal origin isolated from blood between type 2 diabetes and healthy volunteers. | Baseline
  Phosphorylated insulin receptor substrate 1 and its downstream mediators represent the state of neuronal insulin resistance, whose improvement means better insulin signaling. For individuals with type 2 diabetes mellitus and healthy volunteers, blood samples will be collected and stored at -80℃ at baseline. The NEVs isolation and biomarker measurements will be processed uniformly, and the difference of the level of insulin signaling between two groups will be used for exploring underlying mechanism of disease.
The difference of the score of the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery between type 2 diabetes and healthy volunteers. | Baseline
  The cognitive function of interventional participants will be assessed using the Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery. Evaluator convert raw scores to scale scores, then to normalized T scores. T scores of seven domains and composite score are further calculated. The difference of T scores between two groups will be used for evaluating cognitive function. (higher score means better function).
The difference of c-fMRI between type 2 diabetes and healthy volunteers. | Baseline
  The resting-state functional MRI(fMRI) will be conducted at fasting state and after the application of 160 units nasal insulin spray. For every participants, the changes in fMRI (c-fMRI) under the application of nasal insulin spray will be analysed. The c-fMRI between type 2 diabetes and healthy volunteers may reflect the underlying mechanism of disease.

SECONDARY OUTCOMES:
The difference of Diffusion Tensor Imaging scanned by MRI between type 2 diabetes and healthy volunteers | Baseline
  Diffusion Tensor Imaging (DTI) will be performed using diffusion-weighted echo planar imaging sequences. The analysis of DTI will be conducted to investigate the difference of brain structure and morphology between type 2 diabetes and healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, PhD, Principal Investigator — Department of Psychiatry, The Second Xiangya Hospital of Central South University
Locations (1):
- Department of Psychiatry, National Clinical Research Center for Mental Disorders, and National Center for Mental Disorders, The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No